CLINICAL TRIAL: NCT04434794
Title: Treatment of Gingival Recession Using Autologous Adipose-derived Mesenchymal Stem Cells
Brief Title: Treatment of Gingival Recession Using Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(GR2)
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Gingival Recession
Keywords: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): standard treatment according to clinical protocols plus mesenchymal stem cells
  Interventions: Biological: mesenchymal stem cells; Other: standard treatment
- control (Active Comparator): standard treatment according to clinical protocols
  Interventions: Other: standard treatment

INTERVENTIONS:
Biological: mesenchymal stem cells — autologous mesenchymal stem cells
  Arms: mesenchymal stem cells
Other: standard treatment — standard treatment according to clinical protocols

SUMMARY:
Treatment of patients with gingival recession by injection of autologous adipose-derived mesenchymal stem cells mixed with collagen gel

DETAILED DESCRIPTION:
Treatment of patients with gingival recession by injection of autologous adipose-derived mesenchymal stem cells mixed with collagen gel (1×106cells/0.2 ml). The volume of the mixture is divided into 4 equal injections in the gingival region of one tooth (one place injection volume is 0.05 ml of mixture).

ELIGIBILITY:
Inclusion Criteria:

-gingival recession

Exclusion Criteria:

* pregnancy
* breast-feeding
* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
number of patients cured | 1 month
  number of patients cured

CONTACTS AND LOCATIONS:
Overall Officials: Igor D Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Sergey Rubnikovich, Prof, Study Director — Head of the Department of Prosthodontics of BMAPE
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No